CLINICAL TRIAL: NCT02157506
Title: A Phase IIa Study of the Safety, Tolerability and Hemodynamic Effects of a Continuous 6 Hour Intravenous Infusion of CXL-1427 in Hospitalized Patients With Systolic Heart Failure
Brief Title: A Dose Ranging Phase IIa Study of 6 Hour Intravenous Dosages of CXL-1427 in Patients Hospitalized With Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Cardioxyl Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CXL-1427-02; CV013-006 (Other: BMS)
Record Dates: First submitted 2014-05-28; First posted 2014-06-06 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure; Decompensated Heart Failure; Acute Heart Failure
Keywords: Acute Heart failure; Hemodynamics; Pharmacokinetics; Renal Function
MeSH Terms: conditions — Heart Failure | interventions — Glucose; Potassium Acetate; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- CXL-1427 Starting Dose (Experimental): The Starting dose of CXL-1427 in the dose escalation arms will be 3mcg/kg/min
  Interventions: Drug: CXL-1427
- CXL-1427 Dose Level 2 (Experimental): The Second Dose level of CXL-1427 will be evaluated in the Dose Escalation Arm of the study as determined by the independent dose escalation committee
  Interventions: Drug: CXL-1427
- CXL-1427 Dose Level 3 (Experimental): The Third Dose level of CXL-1427 will be evaluated in the Dose Escalation Arm of the study as determined by the independent dose escalation committee
  Interventions: Drug: CXL-1427
- CXL-1427 Dos Level 3 (Experimental): The Third Dose level of CXL-1427 will be evaluated in the Dose Escalation Arm of the study as determined by the independent dose escalation committee
  Interventions: Drug: CXL-1427
- CXL-1427 Dose Level 4 (Experimental): The forth level of CXL-1427 will be evaluated in the Dose Escalation Arm of the study as determined by the independent dose escalation committee
  Interventions: Drug: CXL-1427
- Expansion Cohort 1 (Experimental): Up to 16 Patients will be enrolled across 1 or more of the previously evaluated Dose escalation Levels as determined by the independent dose escalation committee
  Interventions: Drug: CXL-1427
- Placebo for Dose Escalation and Expansion Cohort (Placebo Comparator): Each Dose escalation Arm of the study will have a placebo group in a 2:1 ratio to active treatment for the first 3 patients enrolled and 4:1 to active treatment in the remaining 5 patients so that the overall randomization ratio in each Dose escalation arm will be 3:1 active to placebo. In the expansion Cohort of the study, the ratio of patients randomized to receive a 6-hour infusion of active CXL-1427 or placebo will be 3:1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CXL-1427
  Other Names: BMS-986231
  Arms: CXL-1427 Dos Level 3; CXL-1427 Dose Level 2; CXL-1427 Dose Level 3; CXL-1427 Dose Level 4; CXL-1427 Starting Dose; Expansion Cohort 1
Drug: Placebo
  Other Names: 5% Dextrose & 10mM potassium acetate as same IV solution diluents used in active
  Arms: Placebo for Dose Escalation and Expansion Cohort

SUMMARY:
A randomized, double-blinded, placebo-controlled study of continuous 6-hour IV infusions of CXL-1427 in hospitalized patients with systolic heart failure.

DETAILED DESCRIPTION:
This is a dose finding, randomized, double-blinded, placebo-controlled study of continuous 6-hour IV infusions of CXL-1427 in hospitalized patients with systolic heart failure which will first evaluate up to four ascending dose levels of CXL-1427 in up to four cohorts of 8 patients each (the "Dose Escalation" cohorts). Subsequently, up to three of the initial dose levels of CXL-1427 may be assessed in the additional "Expansion" cohorts of up to approximately 16 patients to gain further confidence in the results at these dose levels. The CXL-1427 dose that will be evaluated in the first cohort will be 3µg/kg/min. The dose levels for the next three sequential Dose Escalation cohorts will be dependent on clinical safety and tolerability, as well as the results of the invasive hemodynamic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria -In order to be eligible for study participation, a patient MUST:
* Be ≥ 18 and ≤ 85 years of age;
* Have a left ventricular ejection fraction (LVEF) ≤40%, as assessed by echocardiography, a multigated acquisition (MUGA) scan or magnetic resonance imaging (MRI) within 3 months prior to or during the current hospitalization;
* Be hospitalized with a primary heart failure or heart failure-related reason, e.g., acute decompensation of heart failure, transplant evaluation, hemodynamic optimization prior to ambulatory inotropes or left ventricular assist device placement;
* Have an indwelling pulmonary artery (PA) catheter in place for assessment of central hemodynamic parameters; [Note: The indwelling catheter may already be in place for medically-indicated reasons, OR be placed for the primary purpose of monitoring the hemodynamic effects of the study drug. If the pulmonary artery catheter is to be placed for the sole purpose of monitoring the hemodynamic effect of the study drug, the patient must have a cardiac index (CI) ≤ 2.2L/min•m2 as measured by a non-invasive cardiac output monitor (NICaS device) ≤6 hours prior to placement of the catheter. In this setting, Exclusion Criteria 3 below also applies.]
* Have a Fick and/or thermodilution determination of cardiac index ≤2.5L/min•m2 at screening, i.e., ≤4 hours before the intended start of the study drug infusion; [Note: For determinations of CI using the thermodilution method, a mean of three consecutive values measured approximately 5 minutes apart, none of which differs from the mean value by more than 15%, should be used.]
* Have a screening and baseline PCWP (or PAD, if a PCWP waveform cannot be reliably obtained) of ≥20 mmHg if systolic blood pressure is ≥100mmHg OR ≥22mmHg if systolic blood pressure is between 95-99mmHg (inclusive);
* Be considered sufficiently stable to be expected not to require administration of any IV or oral vasoactive medications, including diuretics, for at least ~10 hours, i.e., from 4 hours before performing baseline hemodynamic assessments until after the completion of the 6-hour study drug infusion;
* Have a body weight of at least 50kg (110 pounds), but not more than 125kg (275 pounds), and have a body mass index (BMI) <40kg/m2;
* Have adequate peripheral forearm vein access or an available central line port for administration of study drug;
* Be capable of understanding the nature of the trial; be willing and able to comply with the inpatient and outpatient study protocol requirements for the duration of the study (screening period, treatment period, and 30-day post-infusion follow-up period); and be willing to participate in the study, as documented by written informed consent.

Exclusion Criteria- - In order to be eligible for study participation, a patient MUST NOT:

* Have a heart rate <50 or >110 beats per minute (bpm) at baseline;
* Have a screening OR baseline systolic blood pressure (SBP) of >150mmHg or <100mmHg, if PCWP ≥ 20mmHg, but <22mmHg OR <95mmHg, if PCWP ≥ 22mmHg;
* Have tricuspid or pulmonary valve prosthesis or endocarditis, right heart mass, a history of pneumothorax or hemothorax, a bleeding diathesis that would preclude placement of a PAL, or a history of complications from previous pulmonary artery catheter placement, when a pulmonary artery catheter is to be placed solely for the purposes of monitoring the hemodynamic effects of the study drug; In this setting, patients with multiple intracardiac leads and/or left bundle branch block should have such elective pulmonary artery catheter placement performed under radiologic guidance by experienced personnel, e.g. in the cardiac catheterization laboratory. [Note: Other pertinent history, such as trauma, vascular injury or previous surgery should guide selection of the vessel for PAL placement.]
* Have a primary HF etiology attributable to either restrictive/obstructive cardiomyopathy, idiopathic hypertrophic cardiomyopathy (as defined by any wall thickness > 1.8cm) or uncorrected severe valvular disease as defined by AHA/ACC/ESC criteria;
* Have been treated with dopamine, dobutamine, enoximone, nesiritide, nitroglycerine or nitroprusside within 4 hours, or with levosimendan, amrinone or milrinone within 8 hours, prior to performing baseline hemodynamic assessments, or have an anticipated need to be treated with any of these agents before the completion of the 6-hour study drug infusion;
* Be receiving concomitant parenteral therapy with any antiarrhythmic drugs (oral therapy is allowed);
* Be in atrial fibrillation/flutter with an uncontrolled rate (≥100bpm) at the time of randomization; [Note: Patients with a history of A-fib/flutter are eligible, if heart rate is controlled with a ventricular rate not exceeding 100bpm.]
* Have non-sustained ventricular tachycardia (NSVT) of 10 beats or more during any bedside monitoring within 2 hours prior to randomization, or have excessive premature ventricular contractions (PVCs) or complex multifocal ventricular ectopy exceeding 10 beats per minute on a 2-minute rhythm strip taken within 2 hours prior to randomization;
* Require, or be expected to require, any alteration of settings to an implantable cardioverter-defibrillator (ICD), single chamber or biventricular pacemaker, if applicable, from 2 hours before the intended start of the study drug infusion, until after the completion of the study drug infusion;
* Have a history of sudden cardiac death/resuscitation or other appropriate ICD firing within the past 1 year. (Inappropriate ICD firings are not exclusionary);
* Be hospitalized with acute coronary syndrome or acute myocardial infarction during the previous 90 days prior to randomization;
* Have a history of a cerebral vascular accident (CVA or stroke) or of a transient ischemic attack (TIA) within 6 months prior to randomization;
* Have a digoxin level above 1ng/ml (1.281nmol/L) within 8 hours before initiation of the study drug infusion;
* Have persistent abnormal serum electrolytes at baseline, as defined by: a Na+ concentration <130 or >145 mEq/L, or a K+ or Mg2+ concentration outside the normal range (according to the local laboratory); [Note: Any observed electrolyte abnormalities during screening or earlier should be corrected by electrolyte supplementation and within normal acceptable concentrations should be confirmed prior to dosing. Any serum electrolyte abnormalities with associated clinical instability within 8 hours before initiation of the study drug infusion is exclusionary.]
* Have an ALT or AST >3 times the upper normal limit or a hemoglobin <10g/dl (100g/L) within 8 hours before initiation of the study drug infusion;
* Have a serum creatinine >2.5mg/dl (221µmol/L) or severe renal insufficiency [based on any standard limit and equation employed by the local lab, such as a GFR < 30mL/min/1.73m2 according to the Modification of Diet in Renal Disease (MDRD) equation] within 8 hours before initiation of the study drug infusion;
* Have taken an oral phosphodiesterase type 5 inhibitor (PDE5) inhibitor within 96 hours before initiation of the study drug infusion;
* If female, be pregnant or of child-bearing potential (i.e., female patients must be post-menopausal or surgically sterilized);
* Be receiving a drug which is expected to possess a potential for a clinically significant pharmacokinetic interaction with CXL-1427, as defined in the CXL-1427 Investigator's Brochure;
* Be the recipient of a myocardial restraint device or flap;
* Have an anticipated survival of less than 90 days, for any reason;
* Have received an investigational drug, device or biologic product within 30 days (or if longer, 5 half-lives for a drug or biologic agent) prior to randomization, or be planning to receive an investigational agent at any time throughout the full duration of the study until at least 30 days after discontinuation of study drug;
* Have any other clinically significant laboratory abnormality, medical condition or social circumstance that, in the investigator's opinion, makes it inappropriate for the patient to participate in this clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2015-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ShiYin Foo, M.D., Ph D., Study Director — Cardioxyl Pharmaceuticals
Locations (30):
- United States (13):
  - Cardioxyl Study Site, Gainesville, Florida
  - Cardioxyl Study Site, Jacksonville, Florida
  - Cardioxyl Study Site, Macon, Georgia
  - Cardioxyl Study Site, Baltimore, Maryland
  - Cardioxyl Study Site, Detroit, Michigan
  - Cardioxyl Study Site, Newark, New Jersey
  - Cardioxyl Study Site, Chapel Hill, North Carolina
  - Cardioxyl Study Site, Cincinnati, Ohio
  - Cardioxyl Study Site, Columbus, Ohio
  - Cardioxyl Study Site, Charleston, South Carolina
  - Cardioxyl Study Site, Nashville, Tennessee
  - Cardioxyl Study Site, Salt Lake City, Utah
  - Cardioxyl Study Site, Richmond, Virginia
- Germany (7):
  - Cardioxyl Study Site, Bad Neuheim
  - Cardioxyl Study Site, Cologne
  - Cardioxyl Study Site, Frankfurt
  - Cardioxyl Study Site, Göttingen
  - Cardioxyl Study Site, Greifswald
  - Cardioxyl Study Site, Kiel
  - Cardioxyl Study Site, Regensberg
- Jordan (2):
  - Cardioxyl Study Site, Amman
  - Cardioxyl Study Site, Irbid
- Poland (4):
  - Cardioxyl Study Site, Lodz
  - Cardioxyl Study SIte, Warsaw
  - Cardioxyl Study Site, Warsaw
  - Cardioxyl Study Site, Wroclaw
- Russia (4):
  - Cardioxyl Study Site, Kemerovo
  - Cardioxyl Study Site, Moscow
  - Cardioxyl Study Site, Saint Petersburg
  - Cardioxyl Study Site, Tomsk

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 70 participants were enrolled of which only 46 participants received treatment. 24 were not treated due to screen failures, 3 of the 24 were randomized but not dosed due to other reasons.
Groups:
- Placebo: Subjects received matching placebo intravenous (IV) infusion.
- CXL-1427 3μg/kg/Min: Subjects received CXL-1427 3 microgram per kilogram per minute (μg/kg/min) IV infusion as 90 milliliter (mL) of dosing solution at a rate of 15 milliliter per hour (mL/hour) for six hours.
- CXL-1427 5μg/kg/Min: Subjects received CXL-1427 5 μg/kg/min IV infusion as 90 mL of dosing solution at a rate of 15 mL/hour for six hours.
- CXL-1427 7μg/kg/Min: Subjects received CXL-1427 7 μg/kg/min IV infusion as 150 mL of dosing solution at a rate of 25 mL/hour for six hours.
- CXL-1427 12μg/kg/Min: Subjects received CXL-1427 12 μg/kg/min IV infusion as 180 mL of dosing solution at a rate of 30 mL/hour for six hours.
Period: Overall Study
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Started | 12 | 6 | 9 | 12 | 7
Completed | 12 | 5 | 8 | 12 | 7
Not Completed | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min | Total
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.25) | 63.5 (3.51) | 61.1 (11.36) | 61.6 (10.26) | 48.3 (17.49) | 60.0 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 0 | 2 | 7
  Male | 10 | 4 | 8 | 12 | 5 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: A treatment-emergent adverse event (TEAE) was defined as an AE with onset after the start of the study drug infusion at Hour 00:00 through 30 days after the stop of the study drug infusion. All TEAEs and pertinent subsets of TEAEs (e.g., TEAEs with onset during the infusion of study drug, serious TEAEs, etc.) were summarized by system organ class (SOC), preferred term (PT) and treatment group
Time Frame: 30 days following the initiation of treatment
Population: The safety analysis set consists of all randomized participants who received all or part of the infusion of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7
Participants
  At least one TEAE | 3 | 5 | 5 | 7 | 3
  At least one Severe TEAE | 0 | 4 | 0 | 2 | 1
  At least one Drug-related severe TEAE | 0 | 0 | 0 | 0 | 0
  At least one Serious TEAE | 1 | 3 | 1 | 3 | 1
  At least one Drug-related serious TEAE | 0 | 0 | 0 | 0 | 0
  At least one Fatal TEAE | 0 | 1 | 0 | 0 | 0
  At least one Drug-related fatal TEAE | 0 | 0 | 0 | 0 | 0
  At least one TEAE leading to drug interruption | 0 | 0 | 0 | 0 | 0
  At least one TEAE leading to drug discontinuation | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Mean Time Averaged Change From Baseline in Adjudicated Pulmonary Capillary Wedge Pressure (PCWP) During Infusion
Description: The effect of CXL-1427 on PCWP is presented as the mean time-averaged change from baseline over the course of infusion of CXL-1427 or placebo in adjudicated pulmonary capillary wedge pressure (PCWP) on a modified intent-to-treat population
Time Frame: Baseline, Hour 2, Hour 4, Hour 6, Hour 8 post infusion
Population: Modified Intent-To-Treat Analysis Set: all randomized participants who received all or part of the infusion of the study drug and had at least one baseline and post-baseline invasive hemodynamic assessment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7
mm Hg | -0.17 (2.35) | -3.00 (3.06) | -5.06 (3.93) | -4.42 (4.00) | -4.75 (3.50)
Statistical Analysis 1: Comparison: Placebo vs CXL-1427 3μg/kg/Min; Test type: Superiority; p = 0.0059, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 2: Comparison: Placebo vs CXL-1427 5μg/kg/Min; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 3: Comparison: Placebo vs CXL-1427 7μg/kg/Min; Test type: Superiority; p = 0.0062, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 4: Comparison: Placebo vs CXL-1427 12μg/kg/Min; Test type: Superiority; p = 0.0086, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity

3. Primary Outcome: Mean Time-Averaged Change From Baseline in Adjudicated Pulmonary Artery Diastolic Pressure (PAD) During the Infusion
Description: Pulmonary artery diastolic pressure (PAD) was measured by an indwelling PA catheter. Pulmonary artery diastolic pressure (PAD) approximates pulmonary capillary wedge pressure in normal individuals. The effects of CXL-1427 on time-averaged PAD during the course of the infusion are presented.
Time Frame: Baseline, Hour 2, Hour 4, Hour 6, Hour 8 post infusion initiation
Population: Modified Intent-To-Treat Analysis Set: all randomized patients who received all or part of the infusion of the study drug and had at least one baseline and post-baseline invasive hemodynamic assessment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7
mm Hg | -0.21 (3.35) | -3.69 (2.55) | -4.17 (4.02) | -2.67 (3.63) | -3.17 (1.82)
Statistical Analysis 1: Comparison: Placebo vs CXL-1427 3μg/kg/Min; Test type: Superiority; p = 0.0076, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 2: Comparison: Placebo vs CXL-1427 5μg/kg/Min; Test type: Superiority; p = 0.0052, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 3: Comparison: Placebo vs CXL-1427 7μg/kg/Min; Test type: Superiority; p = 0.1064, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 4: Comparison: Placebo vs CXL-1427 12μg/kg/Min; Test type: Superiority; p = 0.1151, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity

4. Primary Outcome: Mean Time-Averaged Percent Change From Baseline in Cardiac Index (Fick)
Description: Cardiac index is a measure of cardiac function, relating the cardiac output from the left ventricle in one minute to body surface area. It is calculated using the Fick principle, using oxygen consumption measured with a metabolic cart, hemoglobin levels, and the difference between arterial and superior vena cava oxygen saturation measured by co-oximetry. Cardiac index as calculated by the Fick method was performed using an assumed oxygen consumption value of 125 ml/min per m2 of body surface area. i.e., an assumed Fick method.
Time Frame: Baseline, Hour 2, Hour 4, Hour 6, Hour 8 post infusion initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7
Percentage of change | 7.95 (16.15) | 0.53 (18.12) | 13.41 (23.53) | 9.59 (11.91) | -9.58 (18.02)
Statistical Analysis 1: Comparison: Placebo vs CXL-1427 3μg/kg/Min; Test type: Superiority; p = 0.4241, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 2: Comparison: Placebo vs CXL-1427 5μg/kg/Min; Test type: Superiority; p = 0.4035, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 3: Comparison: Placebo vs CXL-1427 7μg/kg/Min; Test type: Superiority; p = 0.8308, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 4: Comparison: Placebo vs CXL-1427 12μg/kg/Min; Test type: Superiority; p = 0.1180, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity

5. Secondary Outcome: Mean Time-Averaged Change From Baseline in Adjudicated Pulmonary Artery Systolic Pressure (PAS) During the Infusion
Description: Pulmonary artery systolic pressure (PAS) was measured by an indwelling PA catheter. The effects of CXL-1427 on time-averaged PAS during the course of the infusion are presented
Time Frame: Baseline, Hour 2, Hour 4, Hour 6, Hour 8 post infusion initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7
mm Hg | -0.73 (3.73) | -6.42 (2.59) | -5.98 (5.31) | -6.26 (5.09) | -4.24 (5.24)
Statistical Analysis 1: Comparison: Placebo vs CXL-1427 3μg/kg/Min; Test type: Superiority; p = 0.0048, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 2: Comparison: Placebo vs CXL-1427 5μg/kg/Min; Test type: Superiority; p = 0.0022, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 3: Comparison: Placebo vs CXL-1427 7μg/kg/Min; Test type: Superiority; p = 0.0045, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 4: Comparison: Placebo vs CXL-1427 12μg/kg/Min; Test type: Superiority; p = 0.0294, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity

6. Secondary Outcome: Mean Time-Averaged Change From Baseline in Adjudicated Right Atrial Pressure (RAP) During the Infusion
Description: The effects of CXL-1427 on time-averaged RAP during the course of the infusion are presented
Time Frame: Baseline, Hour 2, Hour 4, Hour 6, Hour 8 post infusion initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7
mm Hg | -0.03 (2.61) | -1.92 (2.91) | -2.08 (3.10) | -2.17 (2.42) | -4.60 (3.23)
Statistical Analysis 1: Comparison: Placebo vs CXL-1427 3μg/kg/Min; Test type: Superiority; p = 0.2022, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 2: Comparison: Placebo vs CXL-1427 5μg/kg/Min; Test type: Superiority; p = 0.0658, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 3: Comparison: Placebo vs CXL-1427 7μg/kg/Min; Test type: Superiority; p = 0.0741, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 4: Comparison: Placebo vs CXL-1427 12μg/kg/Min; Test type: Superiority; p = 0.0497, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity

7. Secondary Outcome: Mean Time-Averaged Change From Baseline in Mean Arterial Blood Pressure (MAP) During the Infusion
Description: Mean arterial pressure during infusion of CXL-1427 or placebo on a modified intent-to-treat population is presented
Time Frame: Baseline, Hour 24 after infusion, Follow-up visit 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7
mm Hg | -1.11 (5.01) | -5.84 (4.46) | -4.75 (10.93) | -7.16 (7.67) | -6.69 (5.67)
Statistical Analysis 1: Comparison: Placebo vs CXL-1427 3μg/kg/Min; Test type: Superiority; p = 0.1842, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 2: Comparison: Placebo vs CXL-1427 5μg/kg/Min; Test type: Superiority; p = 0.3328, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 3: Comparison: Placebo vs CXL-1427 7μg/kg/Min; Test type: Superiority; p = 0.1465, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 4: Comparison: Placebo vs CXL-1427 12μg/kg/Min; Test type: Superiority; p = 0.2799, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity

8. Secondary Outcome: Mean Time-Averaged Change From Baseline in Systolic Blood Pressure (SBP) During the Infusion
Description: Mean Time-Averaged Change from Baseline in Systolic Blood Pressure during infusion of CXL-1427 or placebo on a modified intent-to-treat population is presented
Time Frame: Baseline, Hour 24 after infusion, Follow-up visit 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7
mm Hg | -3.15 (5.53) | -8.69 (4.43) | -2.41 (12.57) | -6.81 (9.54) | -4.64 (4.04)
Statistical Analysis 1: Comparison: Placebo vs CXL-1427 3μg/kg/Min; Test type: Superiority; p = 0.2499, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 2: Comparison: Placebo vs CXL-1427 5μg/kg/Min; Test type: Superiority; p = 0.8281, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 3: Comparison: Placebo vs CXL-1427 7μg/kg/Min; Test type: Superiority; p = 0.4121, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 4: Comparison: Placebo vs CXL-1427 12μg/kg/Min; Test type: Superiority; p = 0.8592, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity

9. Secondary Outcome: Mean Time-Averaged Change From Baseline in Diastolic Blood Pressure (DBP) During the Infusion
Description: Mean Time-Averaged Change from Baseline in Diastolic Blood Pressure during infusion of CXL-1427 or placebo on a modified intent-to-treat population is presented
Time Frame: Baseline, Hour 24 after infusion, Follow-up visit 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7
mm Hg | -0.09 (8.30) | -4.42 (5.22) | -5.93 (11.07) | -7.33 (8.51) | -7.71 (8.03)
Statistical Analysis 1: Comparison: Placebo vs CXL-1427 3μg/kg/Min; Test type: Superiority; p = 0.1391, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 2: Comparison: Placebo vs CXL-1427 5μg/kg/Min; Test type: Superiority; p = 0.1724, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 3: Comparison: Placebo vs CXL-1427 7μg/kg/Min; Test type: Superiority; p = 0.1245, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 4: Comparison: Placebo vs CXL-1427 12μg/kg/Min; Test type: Superiority; p = 0.1690, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity

10. Secondary Outcome: Mean Time-Averaged Change From Baseline in Heart Rate (HR) During the Infusion
Description: Mean Time-Averaged Change from Baseline in Heart Rate during infusion of CXL-1427 or placebo on a modified intent-to-treat population is presented
Time Frame: Baseline, Hour 24 after infusion, Follow-up visit 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Placebo | CXL-1427 3μg/kg/Min | CXL-1427 5μg/kg/Min | CXL-1427 7μg/kg/Min | CXL-1427 12μg/kg/Min
Number analyzed (Participants) | 12 | 6 | 9 | 12 | 7
Beats/min | -0.79 (6.34) | 1.06 (3.74) | -3.09 (6.84) | 1.00 (7.08) | -4.52 (16.92)
Statistical Analysis 1: Comparison: Placebo vs CXL-1427 3μg/kg/Min; Test type: Superiority; p = 0.4936, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 2: Comparison: Placebo vs CXL-1427 5μg/kg/Min; Test type: Superiority; p = 0.9920, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 3: Comparison: Placebo vs CXL-1427 7μg/kg/Min; Test type: Superiority; p = 0.2789, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity
Statistical Analysis 4: Comparison: Placebo vs CXL-1427 12μg/kg/Min; Test type: Superiority; p = 0.9100, Mixed Models Analysis; Statistical significance was defined by a P-value < 0.05. No adjustments were made for multiplicity

ADVERSE EVENTS:
Time Frame: All adverse events were reported from signed of informed consent form through 30 days post final infusion of study drug.
Groups:
- CXL-1427 3 μg/kg/Min: Subjects received CXL-1427 3 microgram per kilogram per minute (μg/kg/min) IV infusion as 90 milliliter (mL) of dosing solution at a rate of 15 milliliter per hour (mL/hour) for six hours.
- CXL-1427 5 μg/kg/Min: Subjects received CXL-1427 5 μg/kg/min IV infusion as 90 mL of dosing solution at a rate of 15 mL/hour for six hours.
- CXL-1427 7 μg/kg/Min: Subjects received CXL-1427 7 μg/kg/min IV infusion as 150 mL of dosing solution at a rate of 25 mL/hour for six hours.
- CXL-1427 12 μg/kg/Min: Subjects received CXL-1427 12 μg/kg/min IV infusion as 180 mL of dosing solution at a rate of 30 mL/hour for six hours.
Arm/Group | Placebo | CXL-1427 3 μg/kg/Min | CXL-1427 5 μg/kg/Min | CXL-1427 7 μg/kg/Min | CXL-1427 12 μg/kg/Min
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/6 | 0/9 | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/12 | 3/6 | 1/9 | 3/12 | 1/7
Other Adverse Events (participants affected / at risk) | 3/12 | 6/6 | 6/9 | 7/12 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | CXL-1427 3 μg/kg/Min (N=6) | CXL-1427 5 μg/kg/Min (N=9) | CXL-1427 7 μg/kg/Min (N=12) | CXL-1427 12 μg/kg/Min (N=7)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | CXL-1427 3 μg/kg/Min (N=6) | CXL-1427 5 μg/kg/Min (N=9) | CXL-1427 7 μg/kg/Min (N=12) | CXL-1427 12 μg/kg/Min (N=7)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.